CLINICAL TRIAL: NCT04531839
Title: Improving the Outcome of Very Preterm Infants Using Evidence-based Collaborative Quality Improvement: A Multi-center Prospective Study
Brief Title: Improving Outcome of Very Preterm Infants Using Collaborative Quality Improvement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SH-EPIQ 20200826
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Morbidity;Newborn; Morality
Keywords: Very preterm infant; Quality improvement; Mortality; Morbidities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention period (Experimental): The 1.5-year period during which all six participating centers receive evidence-based collaborative quality improvement interventions including benchmarking, potential better practice list, PDSA implementation, and collaborative learning
  Interventions: Behavioral: Evidence-based collaborative quality improvement
- Baseline period (No Intervention): The 2-year period before the collaborative quality improvement intervention

INTERVENTIONS:
Behavioral: Evidence-based collaborative quality improvement — Evidence-based collaborative quality improvement interventions including benchmarking, potential better practice list, PDSA implementation and collaborative learning
  Arms: Intervention period

SUMMARY:
A multicenter interventional study using evidence-based collaborative quality improvement to reduce mortality and major morbidities of very preterm infants in six neonatal centers in Shanghai

DETAILED DESCRIPTION:
A multicenter interventional study using evidence-based collaborative quality improvement to reduce mortality and major morbidities of very preterm infants using evidence-based collaborative quality improvement interventions including benchmarking, potential better practice list, PDSA implementation and collaborative learning.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at >=24+0 weeks' gestation and <32+0 weeks' gestation;
2. Admitted to the participating NICUs within 7 days after birth during study period

Exclusion Criteria:

1. Infants with major congenital anomalies;
2. Infants who transferred to non-participating hospitals within 24 hours after birth;

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality or any major morbidity | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if death or with any of the following major morbidities: bronchopulmonary dysplasia, necrotizing stage II or above, retinopathy of prematurity stage III or above, intraventricular hemorrhage grade III or above or cystic periventricular leukomalacia and late-onset epsis

SECONDARY OUTCOMES:
Mortality | During the procedure (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients dead during hospitalization or 28 days after discharge against medical advice
Bronchopulmonary dysplasia | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients reveived respiratory support or oxygen at 36 weeks' corrected gestational age or on discharge
Necrotizing enterocolitis | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients appeared with NEC stage II or above
Severe brain injury | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients appeared with intraventricular hemorrhage grade III or above within 28 days after birth or cystic periventricular leukomalacia
Retinopathy of prematurity | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients appeared with ROP stage III or above.
Late-onset sepsis | During first NICU hospitalization (about 1-4 months)
  It is a binary varibale (1/0). The variabel would be setted into "1",if patients appeared with culture-proven sepsis after 72 hours after birth
Length of NICU stay | During first NICU hospitalization (about 1-4 months)
  days for the first NICU hospitalization

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Obstetrics and Gynecoloy Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hosipital, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Rysavy MA, Li L, Bell EF, Das A, Hintz SR, Stoll BJ, Vohr BR, Carlo WA, Shankaran S, Walsh MC, Tyson JE, Cotten CM, Smith PB, Murray JC, Colaizy TT, Brumbaugh JE, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Between-hospital variation in treatment and outcomes in extremely preterm infants. N Engl J Med. 2015 May 7;372(19):1801-11. doi: 10.1056/NEJMoa1410689. PMID 25946279
- [Background] Smith LK, Blondel B, Van Reempts P, Draper ES, Manktelow BN, Barros H, Cuttini M, Zeitlin J; EPICE Research Group. Variability in the management and outcomes of extremely preterm births across five European countries: a population-based cohort study. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F400-F408. doi: 10.1136/archdischild-2016-312100. Epub 2017 Feb 23. PMID 28232518
- [Background] Soll RF, McGuire W. Evidence-Based Practice: Improving the Quality of Perinatal Care. Neonatology. 2019;116(3):193-198. doi: 10.1159/000496214. Epub 2019 Jun 5. PMID 31167207
- [Background] Zeitlin J, Manktelow BN, Piedvache A, Cuttini M, Boyle E, van Heijst A, Gadzinowski J, Van Reempts P, Huusom L, Weber T, Schmidt S, Barros H, Dillalo D, Toome L, Norman M, Blondel B, Bonet M, Draper ES, Maier RF; EPICE Research Group. Use of evidence based practices to improve survival without severe morbidity for very preterm infants: results from the EPICE population based cohort. BMJ. 2016 Jul 5;354:i2976. doi: 10.1136/bmj.i2976. PMID 27381936
- [Background] Zaka N, Alexander EC, Manikam L, Norman ICF, Akhbari M, Moxon S, Ram PK, Murphy G, English M, Niermeyer S, Pearson L. Quality improvement initiatives for hospitalised small and sick newborns in low- and middle-income countries: a systematic review. Implement Sci. 2018 Jan 25;13(1):20. doi: 10.1186/s13012-018-0712-2. PMID 29370845
- [Background] Zhou Q, Lee SK, Jiang SY, Chen C, Kamaluddeen M, Hu XJ, Wang CQ, Cao Y. Efficacy of an infection control program in reducing ventilator-associated pneumonia in a Chinese neonatal intensive care unit. Am J Infect Control. 2013 Nov;41(11):1059-64. doi: 10.1016/j.ajic.2013.06.007. Epub 2013 Sep 14. PMID 24041863
- [Background] Lee SK, Beltempo M, McMillan DD, Seshia M, Singhal N, Dow K, Aziz K, Piedboeuf B, Shah PS; Evidence-based Practice for Improving Quality Investigators. Outcomes and care practices for preterm infants born at less than 33 weeks' gestation: a quality-improvement study. CMAJ. 2020 Jan 27;192(4):E81-E91. doi: 10.1503/cmaj.190940. PMID 31988152